CLINICAL TRIAL: NCT06989528
Title: Midwifery Students' Opinions on the Process of Preparing Educational Materials in Midwifery Education and Evaluation of the Prepared Materials
Brief Title: Midwifery Students' Opinions on Educational Material Development and Evaluation in Birth Education
Status: Active, not recruiting | Type: Observational
Sponsor: Antalya Bilim University (Other)
Responsible Party: Principal Investigator, Şafak Gür, Master, Antalya Bilim University
Other Study IDs: 2024\992; Antalya Bilim University (Other: Faculty of Health Sciences)
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Educational Problems; Student
Keywords: Midwifery Students; Educational Materials; Maternal Health Education; Postpartum Period

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This qualitative study aims to explore the experiences of midwifery students in preparing educational materials as part of the "Normal Birth and Postpartum Period" course at Antalya Bilim University. The study will evaluate both the students' perspectives on the preparation process and the educational materials they developed. The research is designed to support the development of professional skills by engaging students in the creation of tangible learning tools such as models and visual materials.

DETAILED DESCRIPTION:
The study focuses on evaluating the experiences of third-year midwifery students enrolled in the "Normal Birth and Postpartum Period" course during the 2024-2025 academic year. Participants will be asked to develop educational materials in digital, printed, or physical formats. The materials will be anonymized and evaluated by five experts holding doctoral degrees in midwifery or related fields, using criteria such as scientific accuracy, content depth, visual quality, creativity, usability, and clinical applicability.

Additionally, semi-structured interviews will be conducted with approximately 15-20 voluntary participants to gather in-depth feedback on their experience. The interview data will be analyzed using thematic analysis, while the materials will be assessed via content analysis. Inter-rater reliability among experts will be calculated using Intraclass Correlation Coefficient (ICC).

The study adheres to the Helsinki Declaration, and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* 3rd-year midwifery students
* Enrolled in the "Normal Birth and Postpartum Period" course
* Voluntary participation and informed consent
* Completion of material preparation task

Exclusion Criteria:

* Withdrawal from the course or failure to attend data collection sessions
* Incomplete or substandard educational material submission

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Third-year midwifery students enrolled in the "Normal Birth and Postpartum Period" course at Antalya Bilim University during the 2024-2025 academic year. Participants are selected from a total of 39 students based on voluntary participation and willingness to complete the educational material preparation process.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Themes identified in students' responses during semi-structured interviews on the impact of educational material preparation on professional knowledge and skills | January 2025 (end of the course)
  Qualitative data will be collected via semi-structured interviews conducted with 15-20 midwifery students at the end of the course. Thematic analysis will be performed to identify recurring themes related to knowledge acquisition, skill development, motivation, problem-solving, and integration of theory into practice. Interviews will be audio-recorded, transcribed, and coded by at least two independent researchers to ensure reliability.
Scores assigned to educational materials prepared by students, based on expert rubric assessing scientific accuracy, usability, visual quality, and clinical applicability | December 2024 - January 2025 (evaluation phase)
  Five faculty experts with doctoral-level qualifications will evaluate each student-created educational material using a standardized scoring rubric with 7 criteria. Each criterion will be scored on a 5-point Likert scale (1 = poor, 5 = excellent). Total score range: 7-35. Higher scores indicate better quality and relevance. Inter-rater reliability will be assessed using the Intraclass Correlation Coefficient (ICC). The materials will be anonymized and scored independently.

SECONDARY OUTCOMES:
Themes identified in students' suggestions for improving the educational material preparation process in midwifery education | At the end of the course (May 2025)
  Qualitative data will be gathered through semi-structured interviews conducted at the end of the course. Students will be asked open-ended questions regarding their suggestions for improving the process of creating educational materials. Interviews will be transcribed and thematically analyzed to extract recurring suggestions and improvement areas related to instructional design, time management, group work, access to resources, and integration with clinical learning. Two independent researchers will code the data, and discrepancies will be resolved by consensus.
Themes identified in students' experiences related to motivation and professional development during the educational material preparation process | At the end of the course (May 2025)
  Semi-structured interviews will be conducted with 15-20 midwifery students at the end of the course. Students will reflect on how the process of developing educational materials affected their motivation, self-efficacy, and sense of professional identity. Thematic analysis will be used to identify key themes such as increased confidence, engagement, sense of responsibility, and future professional aspirations. Interviews will be coded independently by two researchers to ensure analytical reliability.
Themes identified in students' perceptions of digital skill development and technology use during the educational material preparation process | At the end of the course (May 2025)
  Through semi-structured interviews, students will be asked to evaluate how the material development process contributed to their ability to use digital tools (e.g., presentation software, graphic design platforms, video creation tools). Thematic analysis will identify perceived improvements in digital literacy, confidence in using educational technology, and barriers experienced. Coding will be performed using qualitative analysis software and reviewed by multiple researchers for consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Serhatlıoğlu, Döşemealtı, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study is qualitative, and the data include semi-structured interview transcripts and student-created educational materials.
  Even though materials are anonymized, sharing detailed qualitative data could still pose confidentiality and ethical concerns, especially in a small student population.
  No biospecimens or numeric datasets are involved.